CLINICAL TRIAL: NCT07388238
Title: Ultrasound Guided Pectoral Nerve Block (PEC I) Versus Serratus Anterior Plane Block (SAPB) for Postoperative Analgesia in Modified Radical Mastectomy
Brief Title: Ultrasound-Guided PEC I vs SAP Block for Postoperative Analgesia in Modified Radical Mastectomy
Acronym: PECS I vs SAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mariam Kamal Habib, Principal investigatir, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MS 263/ 2021
Record Dates: First submitted 2026-01-26; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Modified Radical Mastectomy; Pectoral Nerve Blocks; Serratus Anterior Plane Block
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This study follows a randomized parallel-group interventional model comparing two established regional anesthesia techniques: PEC block and SAP block. Participants are randomly allocated in a 1:1 ratio using concealed assignment to ensure unbiased group distribution. Each participant receives only the technique assigned, with no crossover permitted. Standardized protocols are applied for induction, drug dosing, positioning, and monitoring to minimize procedural variability. Outcome assessors and data collectors are blinded to group allocation whenever feasible. Both groups follow identical perioperative timelines, including preoperative evaluation, intraoperative monitoring, and postoperative pain assessment. This model allows a controlled and unbiased comparison of the efficacy, safety, and clinical performance of the two techniques under uniform conditions.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-Guided Pectoral Nerve Block (PECS I) Arm (Experimental): Participants in this arm receive an ultrasound-guided pectoral nerve block (PECS I) after induction of general anesthesia, using 20 mL of 0.25% bupivacaine injected into the interpectoral plane between the pectoralis major and pectoralis minor muscles for postoperative analgesia following modified radical mastectomy.
  Interventions: Procedure: Ultrasound-Guided Pectoral Nerve Block (PECS I)
- Ultrasound-Guided Serratus Anterior Plane Block (SAPB) Arm (Experimental): Participants in this arm receive an ultrasound-guided serratus anterior plane block after induction of general anesthesia, using 20 mL of 0.25% bupivacaine injected between the serratus anterior muscle and the external intercostal muscles for postoperative analgesia following modified radical mastectomy.
  Interventions: Procedure: Ultrasound-Guided Serratus Anterior Plane Block (SAPB)

INTERVENTIONS:
Procedure: Ultrasound-Guided Pectoral Nerve Block (PECS I) — Participants receive an ultrasound-guided pectoral nerve block (PECS I) after induction of general anesthesia. A 20 mL solution of 0.25% bupivacaine is injected into the interpectoral plane between the pectoralis major and minor muscles. The block is performed under aseptic conditions using an in-plane needle approach from medial to lateral for postoperative analgesia following modified radical mastectomy.
  Arms: Ultrasound-Guided Pectoral Nerve Block (PECS I) Arm
Procedure: Ultrasound-Guided Serratus Anterior Plane Block (SAPB) — Participants receive an ultrasound-guided serratus anterior plane block after induction of general anesthesia. A 20 mL solution of 0.25% bupivacaine is injected between the serratus anterior muscle and the external intercostal muscles at the midaxillary line under aseptic conditions. The block is performed using an in-plane needle approach from caudal to cranial for postoperative analgesia following modified radical mastectomy.
  Arms: Ultrasound-Guided Serratus Anterior Plane Block (SAPB) Arm

SUMMARY:
This randomized double-blind controlled clinical trial was conducted to compare the analgesic efficacy of ultrasound-guided Pectoral Nerve Block versus Serratus Anterior Plane Block in female patients undergoing Modified Radical Mastectomy. Sixty-four ASA I-II female patients aged 35-60 years were randomly allocated into two equal groups: Group I received PEC I block and Group II received SAPB, using 20 ml of 0.25% bupivacaine in both groups after induction of general anesthesia.

Postoperative pain was assessed using the Numeric Rating Scale (NRS) for 24 hours. Hemodynamic parameters, time to first rescue analgesia, total postoperative opioid consumption, and side effects were recorded. The SAPB group showed significantly lower postoperative pain scores during the first 6 hours, significantly longer time to first rescue analgesia, and significantly lower total pethidine consumption compared to the PEC I group. In addition, mean arterial blood pressure and heart rate were significantly lower intraoperatively and during early postoperative periods in the SAPB group. The incidence of postoperative nausea and vomiting was significantly higher in the PEC I group.

Conclusion: Ultrasound-guided Serratus Anterior Plane Block provides superior postoperative analgesia with better hemodynamic stability and fewer opioid-related side effects compared to Pectoral Nerve Block in patients undergoing Modified Radical Mastectomy

modified radical mastectomy

DETAILED DESCRIPTION:
Postoperative pain following modified radical mastectomy (MRM) is often moderate to severe and may negatively affect patient recovery, increase opioid consumption, and contribute to postoperative complications such as nausea, vomiting, and hemodynamic instability. Regional analgesic techniques have become an integral component of multimodal analgesia strategies aiming to improve pain control while minimizing opioid-related adverse effects. Among these techniques, ultrasound-guided Pectoral Nerve Block (PEC I ) and Serratus Anterior Plane Block (SAPB) have gained increasing attention for breast surgeries. This randomized double-blind controlled clinical trial was designed to compare the efficacy of ultrasound-guided PEC I block versus ultrasound-guided SAPB for postoperative analgesia in female patients undergoing modified radical mastectomy under general anesthesia.

After obtaining approval from the Research Ethics Committee of the Faculty of Medicine, Ain Shams University, and written informed consent from all participants, a total of 64 female patients aged 35-60 years with ASA physical status I or II scheduled for MRM were enrolled. Patients were randomly allocated into two equal groups (32 patients each) using a computer-generated randomization sequence with sealed opaque envelopes to ensure allocation concealment. All patients received standardized general anesthesia. Following induction of anesthesia and under complete aseptic precautions, the assigned regional block was performed using ultrasound guidance. Patients in Group I received an ultrasound-guided PEC I block, where 20 ml of 0.25% bupivacaine was injected into the interpectoral plane between the pectoralis major and pectoralis minor muscles. Patients in Group II received an ultrasound-guided serratus anterior plane block, with 20 ml of 0.25% bupivacaine injected between the serratus anterior muscle and the external intercostal muscles. Postoperative pain intensity was assessed using the Numeric Rating Scale (NRS) for 24 hours. Hemodynamic parameters including heart rate and mean arterial blood pressure were recorded intraoperatively and postoperatively at predefined intervals. The results demonstrated that SAPB provided superior postoperative analgesia compared to PEC I block. Patients in the SAPB group experienced significantly lower pain scores during the first 6 postoperative hours, a significantly longer time to first rescue analgesia, and a significant reduction in total postoperative pethidine consumption. Furthermore, the SAPB group showed better hemodynamic stability during intraoperative and early postoperative periods, with significantly lower heart rate and mean arterial blood pressure. The incidence of postoperative nausea and vomiting was significantly higher in the PEC I group. These findings suggest that ultrasound-guided serratus anterior plane block is a more effective and safer regional analgesic technique than pectoral nerve block for postoperative pain management in patients undergoing modified radical mastectomy, offering improved analgesia, reduced opioid requirements, and fewer adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Physical status: ASA grades I and II
* Age between 35 and 60.

Exclusion Criteria

* Known Allergy to one of the study drugs.
* Pregnant patients.
* Other Malignancy.
* History or evidence of coagulopathy, use of anti coagulant or anti platelet therapy

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 32 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2021-11-06 (Actual); Study Completion 2021-12-09 (Actual)

PRIMARY OUTCOMES:
Postoperative pain intensity measured by Numeric Rating Score (NRS) | Within the first 24 hours postoperatively
  Pain intensity will be assessed using the 10-point NRS at multiple time points: At the entry to the PACU, and at 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 18, 20, 22 and 24 hours postoperatively. NRS scoring: 0 = no pain, 1-3 = mild pain, 4-6= moderate pain, 7-10 = severe pain. The mean NRS score during the first 24 postoperative hours will serve as the primary outcome to evaluate analgesic efficacy between study groups.

SECONDARY OUTCOMES:
Time to first rescue analgesia | From the end of surgery to the administration of the first rescue analgesic.
  The duration in minutes from the end of surgery to the administration of the first rescue analgesic (Diclofenac 75 mg) will be recorded.
Total pethidine consumption after surgery | Within the first 24 hours postoperatively
  The total amount of pethidine (mg) administered to each patient as rescue analgesia during the first 24 hours postoperatively will be recorded. This outcome evaluates the overall analgesic requirement and opioid-sparing effect of the blocks interventions.
Mean arterial blood pressure | Within the first 24 hours postoperatively
  Mean arterial blood pressure (MAP), measured in mmHg, Measurements will be obtained at skin incision, 20min, 40 min and at 60 min intraoperatively then at at 1, 2, 4, 6, 8, 12, 18, and 24 hours postoperatively.
Heart Rate | From the skin incision and up to 24 hours postoperatively
  Heart Rate (HR), measured in (Beat/minute). Measurements will be obtained at skin incision, 20min, 40 min and at 60 min intraoperatively then at at 1, 2, 4, 6, 8, 12, 18, and 24 hours postoperatively.
Adverse events | Within the first 24 hours postoperatively
  Nausea, Vomiting

CONTACTS AND LOCATIONS:
Locations (1):
- Anaethesia Department, Ain Shams University Hospital, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) from this study, including clinical parameters, and demographic information, will be shared with qualified researchers upon request after publication of the study results. Requests will be reviewed by the Principal Investigator, and approved data will be shared via a secure repository. No personal identifiers will be included to ensure participant confidentiality.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Upon publication of the study results.*End Date: 5 years after publication.
Access Criteria: Qualified researchers may request access to de-identified individual participant data (IPD) from this study, including clinical parameters, ventilatory settings, oxygenation indices, and demographic information. Supporting information such as Study Protocol, Statistical Analysis Plan (SAP), and Clinical Study Report (CSR) will also be provided. Requests will be submitted to the Principal Investigator for review. Approved requests will receive the data through a secure repository to ensure confidentiality. Data will not include any personal identifiers, and access is limited to research purposes only.